CLINICAL TRIAL: NCT03085836
Title: An Open-Label, Single-center, Parallel, Phase 1 Study to Determine the Pharmacokinetics of Single- and Multiple- Oral Doses of TAK-438 10 mg and 20 mg in Healthy Adult Chinese Subjects
Brief Title: A Pharmacokinetic Study of TAK-438 in Healthy Adult Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-438_114; U1111-1191-6949 (Registry Identifier: WHO); CTR20170137 (Registry Identifier: CFDA)
Record Dates: First submitted 2017-03-16; First posted 2017-03-21 (Actual); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-08

CONDITIONS: Healthy Participants
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAK-438 10 milligram (mg) Once Daily (Experimental): TAK-438 10 mg, tablets, orally, once daily on Days 1, 3-9. Participants were required to fast for a minimum of 10 hours prior administration of assigned treatment.
  Interventions: Drug: TAK-438
- TAK-438 20 mg Once Daily (Experimental): TAK-438 20 mg, tablets, orally, once daily on Days 1, 3-9. Participants were asked to fast for a minimum of 10 hours prior administration of assigned treatment.
  Interventions: Drug: TAK-438
- TAK-438 20 mg Twice Daily (Experimental): TAK-438 20 mg, tablets, orally, once on Day 1 and twice daily on Days 3-9. Participants were asked to fast for a minimum of 10 hours prior to breakfast, followed by administration of assigned treatment 0.5 hours after breakfast and dinner.
  Interventions: Drug: TAK-438

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets.

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (PK) of TAK-438 in healthy adult Chinese participants after both single and multiple dose administration.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 is being tested in healthy participants in order to evaluate the PK of single and multiple oral dose.

The study will enroll approximately 36 healthy participants. Participants will be assigned to one of the three treatment groups:

* TAK-438 10 mg tablet once daily
* TAK-438 20 mg tablet once daily
* TAK-438 20 mg tablet twice daily All participants will be asked to take TAK-438 tablet at the same time on Day 1 and Days 3-9.

This single-centre trial will be conducted in China. The overall time to participate in this study is 18 days. Participants will remain confined to the clinic from Day 1 up to Day 11 and will be followed-up by telephone or visit on Day 18.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male or female Chinese participant.
2. Is aged 18 to 45 years, inclusive, at the time of signing the informed consent form.
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) between 19 and 26 kilogram per square meter (kg/m^2), inclusive at Screening (Check-In Day -1).
4. Is willing to abstain from caffeine and alcohol from 72 hours before first dose (Day 1) until the Follow-up Visit on Day 18.
5. Is willing to abstain from strenuous exercise from 72 hours before first dose (Day 1) until the Follow-up Visit on Day 18.
6. Is willing to provide a sample for pharmacogenetic analysis (for cytochrome [CYP2C19] genotyping).

Exclusion Criteria:

1. Has uncontrolled, clinically significant cardiovascular disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
2. Is lactose intolerant or has a known hypersensitivity to any component of the formulation of TAK-438.
3. Has poor peripheral venous access.
4. Has donated or lost 400 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to Day 1; or participant has donated or lost more than 200 mL or more of his or her blood in the last 28 days.
5. Has a history of symptomatic gastroesophageal reflux disease (GERD), Erosive Esophagitis, duodenal ulcer (DU), gastric ulcer (GU), dyspepsia, Barrett's Esophagus, or Zollinger-Ellison (ZE) syndrome or has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in China from 19 April 2017 to 17 August 2017.
Pre-assignment Details: Healthy Chinese participants were enrolled in this study to receive treatment in one of the 3 treatment groups: TAK-438 10 milligram (mg) once daily or TAK-438 20 mg once daily or TAK-438-20 mg twice daily.
Groups:
- TAK-438 10 mg Once Daily: TAK-438 10 mg, tablet, orally, once daily on Days 1, 3 to 9. Participants were required to fast for a minimum of 10 hours prior administration of assigned treatment.
- TAK-438 20 mg Once Daily: TAK-438 20 mg, tablet, orally, once daily on Days 1, 3 to 9. Participants were required to fast for a minimum of 10 hours prior administration of assigned treatment.
- TAK-438 20 mg Twice Daily: TAK-438 20 mg, tablet, orally, twice daily on Days 1, 3 to 9. Participants were required to fast for a minimum of 10 hours prior to breakfast, followed by administration of assigned treatment 0.5 hours after breakfast and dinner.
Period: Overall Study
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Started | 12 | 11 | 10
Completed | 12 | 11 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic (PK) set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily | Total
Number analyzed (Participants) | 12 | 11 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  years | 25.2 (2.95) | 23.9 (3.99) | 27.2 (4.83) | 25.4 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    Female | 6 | 5 | 4 | 15
    Male | 6 | 6 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 12 | 11 | 10 | 33
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    China | 12 | 11 | 10 | 33
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  centimeter (cm) | 166.35 (8.426) | 169.59 (7.672) | 164.31 (9.377) | 166.81 (8.498)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  kilogram (kg) | 62.63 (7.601) | 66.05 (8.501) | 61.66 (6.449) | 63.47 (7.597)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  kilogram per square meter (kg/m^2) | 22.63 (2.086) | 22.89 (1.711) | 22.88 (2.110) | 22.79 (1.918)
Smoking classification [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    Never smoked | 12 | 11 | 10 | 33
Alcohol consumption [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    Never drank | 12 | 11 | 10 | 33
Caffeine consumption [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    Had no caffeine consumption | 12 | 11 | 10 | 33
Cytochrome P450 2C19 (CYP2C19) Genotype [Count of Participants; unit: Participants] — Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
  Participants
    *1/*1 | 5 | 4 | 4 | 13
    *1/*2 | 4 | 6 | 5 | 15
    *1/*3 | 1 | 0 | 0 | 1
    *2/*2 | 1 | 1 | 0 | 2
    *2/*3 | 1 | 0 | 1 | 2
    *3/*3 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Free Base of TAK-438 (TAK-438F) and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
nanogram per milliliter (ng/mL)
  TAK-438F | 9.148 (2.9972) | 18.18 (4.4973) | 25.23 (10.017)
  M-I | 38.32 (8.6143) | 67.95 (23.388) | 59.02 (18.443)
  M-II | 2.840 (1.0442) | 5.155 (2.7868) | 4.879 (2.2426)
  M-III | 15.42 (3.7788) | 25.63 (7.8650) | 25.67 (5.9219)
  M-IV-Sul | 28.29 (5.0563) | 60.67 (16.499) | 42.28 (9.1174)

2. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
hour
  TAK-438F | 1.750 [1.00 to 4.02] | 2.000 [0.750 to 4.00] | 2.500 [0.750 to 4.00]
  M-I | 1.500 [0.750 to 2.00] | 1.500 [0.750 to 3.00] | 2.000 [1.00 to 4.00]
  M-II | 4.010 [3.00 to 10.0] | 6.000 [3.00 to 10.0] | 10.00 [3.00 to 12.0]
  M-III | 1.750 [1.00 to 2.00] | 2.000 [1.50 to 3.00] | 2.000 [1.50 to 4.00]
  M-IV-Sul | 1.500 [1.00 to 2.00] | 1.500 [1.50 to 3.00] | 2.000 [1.50 to 3.00]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
hour*nanogram per milliliter (h*ng/mL)
  TAK-438F | 84.38 (29.197) | 188.1 (43.066) | 226.8 (67.128)
  M-I | 305.7 (88.227) | 617.2 (213.56) | 578.7 (144.15)
  M-II | 52.97 (22.843) | 106.3 (74.306) | 117.8 (41.170)
  M-III | 92.83 (34.769) | 178.7 (64.779) | 193.7 (56.808)
  M-IV-Sul | 132.5 (44.602) | 307.5 (89.884) | 240.8 (82.555)

4. Primary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Tau Over the Dosing Interval for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
h*ng/mL
  TAK-438F | 74.91 (24.835) | 168.6 (37.455) | 154.8 (38.920)
  M-I | 251.4 (77.758) | 528.8 (182.62) | 344.1 (91.089)
  M-II | 31.77 (18.646) | 79.07 (56.206) | 41.55 (19.189)
  M-III | 87.98 (31.136) | 169.2 (59.474) | 149.1 (36.714)
  M-IV-Sul | 127.1 (43.648) | 296.0 (86.359) | 192.8 (57.176)

5. Primary Outcome: T1/2z: Terminal Disposition Half-life for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: The PK set included all participants who received the study drug, had sufficient plasma/urine concentration data to calculate at least 1 PK parameter, and completed the minimum protocol specified procedures with no significant protocol deviations. PK analysis population where data at specified time points were available.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
hour
  TAK-438F | 7.879 (1.2352) | 6.996 (1.0110) | 7.116 (0.71638)
  M-I | 10.82 (4.0923) | 8.256 (1.2964) | 8.385 (0.73316)
  M-II: number analyzed (Participants) | 11 | 11 | 8
  M-II | 10.52 (4.3311) | 10.37 (2.9973) | 12.29 (4.0538)
  M-III | 6.695 (1.3786) | 6.335 (1.1833) | 6.791 (0.89228)
  M-IV-Sul | 4.753 (2.4430) | 5.698 (1.2625) | 5.521 (2.2225)

6. Primary Outcome: Cmax,ss: Maximum Observed Plasma Concentration, at Steady State for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: Day 9 pre-dose and at multiple timepoints (up to 24 hours for TAK-483 10 mg once daily and 20 mg once daily; up to 12 hours for TAK-438 20 mg twice daily) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
ng/mL
  TAK-438F | 11.01 (3.4863) | 23.43 (6.1433) | 37.88 (10.910)
  M-I | 43.39 (9.6528) | 79.85 (22.119) | 59.55 (15.512)
  M-II | 3.558 (1.4983) | 6.554 (2.6078) | 9.174 (2.8376)
  M-III | 16.62 (4.1919) | 30.15 (7.3228) | 33.01 (6.1638)
  M-IV-Sul | 25.33 (3.6619) | 54.08 (13.927) | 39.74 (7.1405)

7. Primary Outcome: Tmax, ss: Time to Reach the Maximum Plasma Concentration (Cmax) at Steady State for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
hour
  TAK-438F | 1.500 [0.750 to 3.02] | 2.000 [0.750 to 3.00] | 3.000 [0.750 to 4.00]
  M-I | 1.500 [0.750 to 2.02] | 1.000 [0.750 to 2.00] | 2.500 [1.00 to 10.0]
  M-II | 4.000 [3.00 to 6.00] | 3.000 [3.00 to 10.0] | 3.500 [0.00 to 10.0]
  M-III | 1.750 [1.00 to 3.00] | 2.000 [1.50 to 3.00] | 3.000 [1.50 to 4.00]
  M-IV-Sul | 2.000 [1.00 to 3.00] | 1.500 [1.50 to 2.00] | 3.000 [1.50 to 4.00]

8. Primary Outcome: AUCτ,ss: Area Under the Plasma Concentration-time Curve During a Dosing Interval, at Steady State for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
h*ng/mL
  TAK-438F | 93.90 (28.053) | 212.7 (57.214) | 273.4 (71.830)
  M-I: number analyzed (Participants) | 12 | 11 | 9
  M-I | 285.5 (77.884) | 581.1 (198.14) | 435.3 (92.064)
  M-II: number analyzed (Participants) | 12 | 11 | 7
  M-II | 46.31 (24.298) | 105.5 (51.688) | 100.4 (27.966)
  M-III | 95.94 (29.719) | 194.6 (53.749) | 222.6 (49.670)
  M-IV-Sul | 117.1 (37.489) | 256.1 (62.786) | 225.7 (52.675)

9. Primary Outcome: Aet: Total Amount of Drug Excreted in Urine From Time 0 to Time T for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
microgram (mcg)
  TAK-438F | 448.5 (159.06) | 890.3 (243.24) | 1478 (405.32)
  M-I | 176.6 (79.813) | 253.1 (118.69) | 211.2 (124.21)
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.5120 (1.6191)
  M-IV-Sul | 205.4 (61.587) | 422.1 (143.24) | 387.1 (142.06)

10. Primary Outcome: Fe,t: Fraction of Drug Excreted in Urine From Time 0 to Time t for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
percentage of drug
  TAK-438F | 4.485 (1.5906) | 4.448 (1.2093) | 7.399 (2.0335)
  M-I | 1.760 (0.79678) | 1.262 (0.59122) | 1.053 (0.61992)
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.002460 (0.0077792)
  M-IV-Sul | 1.609 (0.48258) | 1.650 (0.56108) | 1.513 (0.55536)

11. Primary Outcome: CLr: Renal Clearance for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 1
Time Frame: Day 1 pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
liter per hour (L/h)
  TAK-438F | 5.443 (1.0398) | 4.922 (1.4362) | 6.733 (1.3109)
  M-I | 0.6235 (0.16437) | 0.4465 (0.24193) | 0.3753 (0.19679)
  M-II: number analyzed (Participants) | 11 | 11 | 8
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.001820 (0.0057553)
  M-IV-Sul | 1.748 (0.65948) | 1.527 (0.77444) | 1.707 (0.47416)

12. Primary Outcome: Aeτ: Amount of Drug Excreted in Urine During a Dosing Interval for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
mcg
  TAK-438F | 437.7 (121.93) | 859.9 (155.66) | 1327 (274.04)
  M-I | 224.3 (79.531) | 354.1 (165.88) | 340.9 (181.71)
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 205.2 (52.172) | 390.7 (99.477) | 446.4 (139.39)

13. Primary Outcome: Fe,τ: Fraction of Administered Dose of Drug Excreted in Urine During a Dosing Interval for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of drug
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
percentage of drug
  TAK-438F | 4.377 (1.2193) | 4.299 (0.77678) | 6.634 (1.3737)
  M-I | 2.236 (0.79323) | 1.765 (0.82755) | 1.700 (0.90664)
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 1.605 (0.40853) | 1.528 (0.38946) | 1.748 (0.54499)

14. Primary Outcome: CLR: Renal Clearance for TAK-438F and Its Metabolites M-I, M-II, M-III and M-IV-Sul on Day 9
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
Number analyzed (Participants) | 12 | 11 | 10
L/h
  TAK-438F | 4.848 (1.2372) | 4.251 (1.1565) | 4.977 (0.71952)
  M-I: number analyzed (Participants) | 12 | 11 | 9
  M-I | 0.8126 (0.26393) | 0.6207 (0.22632) | 0.7943 (0.39001)
  M-II: number analyzed (Participants) | 12 | 11 | 7
  M-II | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-III | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  M-IV-Sul | 1.931 (0.79907) | 1.614 (0.58643) | 2.067 (0.70761)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to follow-up (Day 1 up to Day 18)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-438 10 mg Once Daily | TAK-438 20 mg Once Daily | TAK-438 20 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 4/12 | 6/11 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-438 10 mg Once Daily (N=12) | TAK-438 20 mg Once Daily (N=11) | TAK-438 20 mg Twice Daily (N=10)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 2 | 2
Red blood cells urine positive (Investigations) | 2 | 0 | 2
Neutrophil count increased (Investigations) | 1 | 1 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT03085836/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT03085836/SAP_001.pdf